CLINICAL TRIAL: NCT06409091
Title: Short Term Outcomes of Heavy-weight Versus Medium-weight Synthetic Mesh in a Retrospective Cohort of Clean-Contaminated and Contaminated Retromuscular Ventral Hernia Repairs
Brief Title: Short Term Outcomes of Heavy-weight Versus Medium-weight Synthetic Mesh
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Lucas Beffa, Assistant Professor of Surgery, The Cleveland Clinic
Other Study IDs: 23-346
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Hernia, Ventral; Hernia Incisional
MeSH Terms: conditions — Hernia, Ventral; Incisional Hernia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Medium weight PP mesh: Patients receiving medium weight PP mesh in clean-contaminated and contaminated settings
  Interventions: Device: Medium weight or Heavy weight mesh
- Heavy Weight PP Mesh: Patients receiving heavy weight PP mesh in clean-contaminated and contaminated settings
  Interventions: Device: Medium weight or Heavy weight mesh

INTERVENTIONS:
Device: Medium weight or Heavy weight mesh — Patients received a hernia repair with one of the two groups

SUMMARY:
This study compares short term outcomes of patients undergoing a hernia repair with heavy weight mesh vs medium weight mesh in clean-contaminated and contaminated cases.

DETAILED DESCRIPTION:
The Abdominal Core Health Quality Collaborative was queried for patients undergoing open retromuscular hernia repairs with both heavy weight polypropylene (PP) mesh and medium weight PP mesh in cases where there was clean-contaminated and contaminated surgeries. The short term outcomes were then evaluated including wound infections, readmissions, recurrences of the hernia, and quality of life scores.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing open ventral hernia repairs with synthetic mesh in contaminated and clean contaminated surgery

Exclusion Criteria:

* Laparoscopic or robotic surgery
* clean cases or dirty cases
* pregnancy
* under age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who underwent open ventral hernia repairs with synthetic mesh in contaminated and clean-contaminated hernia repair surgeries.
Sampling Method: Non-Probability Sample
Enrollment: 1496 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Wound complications | 30 days post op
  Wound complcations

SECONDARY OUTCOMES:
Mesh removal | 30 days post op
  mesh removal after surgery
Readmissions | 30 days post op
  readmission or ER visit after surgery
Reoperations | 30 days post op
  Reoperation after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
This data will not be shared with other researchers other than through peer-reviewed publication